CLINICAL TRIAL: NCT05041725
Title: The Impact of Remimazolam on the Left Ventricular Systolic Performance for Cardiac Surgery: a Speckle Tracking Analysis of the Left Ventricular Strain Using Transthoracic Echocardiography
Brief Title: The Impact of Remimazolam for Postoperative Sedation on the Left Ventricular Systolic Performance in Cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor, Department of Anesthesiology, Konkuk University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210000-2
Record Dates: First submitted 2021-08-31; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — remimazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- remimazolam infusion (Experimental): Intraoperative remimazolam infusion for postoperative sedation
  Interventions: Drug: Remimazolam Injection [Byfavo]

INTERVENTIONS:
Drug: Remimazolam Injection [Byfavo] — Remimazolam injection and continuous infusion for postoperative sedation, 0.2 mg/kg for 1 min and continuous infusion of 1-2 mg/kg/hour
  Other Names: Remimazolam infusion

SUMMARY:
This study analyzes the impact of intraoperative Remimazolam infusion for postoperative sedation on the left ventricular global longitude strain (LV-GLS) patients undergoing cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* elective off-pump coronary artery bypass surgery

Exclusion Criteria:

* arrhythmia
* LV ejection fraction < 50 %
* preoperative inotropic support

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
change of the left ventricular global longitudinal strain | 1 minutes
  mean values of the left ventricular global longitudinal strain after 3 minutes, 5 minutes and 10 minutes after the Remimazolam administration

IPD SHARING:
Plan to Share IPD: No